CLINICAL TRIAL: NCT02411786
Title: A Phase I Study of a DNA Vaccine Encoding Androgen Receptor Ligand-Binding Domain (AR LBD), With or Without Granulocyte Macrophage Colony-Stimulating Factor Adjuvant, in Patients With Metastatic Prostate Cancer
Brief Title: A Phase I Study of a DNA Vaccine Encoding Androgen Receptor Ligand-Binding Domain (AR LBD) +/-GMCSF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Madison Vaccines Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW14072; 2014-1456 (Registry Identifier: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison); NCI-2015-00808 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2015-03-27; First posted 2015-04-08 (Estimated); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; regramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- pTVG-AR biweekly (Experimental): pTVG-AR (dose: 100 µg) alone without rhGM-CSF. Administered at weeks 0, 2, 4, 6, 8, and 10 (biweekly) for 6 doses, then administered at week 12, week 24, week 36, and week 48 (quarterly) for 4 doses, or 10 total doses.
  Interventions: Biological: pTVG-AR
- pTVG-AR staggered biweekly (Experimental): pTVG-AR (dose: 100 µg) alone without rhGM-CSF. Administered at weeks 0, 2, 12, 14, 24, 26, 36, 38, 48 and 50 (staggered biweekly schedule) for 10 total doses.
  Interventions: Biological: pTVG-AR
- pTVG-AR with rhGM-CSF biweekly (Experimental): pTVG-AR (dose: 100 µg) with rhGM-CSF (200 µg). Administered at weeks 0, 2, 4, 6, 8, and 10 (biweekly) for 6 doses, then administered at week 12, week 24, week 36, and week 48 (quarterly) for 4 doses, or 10 total doses.
  Interventions: Biological: pTVG-AR; Biological: gm-csf
- pTVG-AR with rhGM-CSF staggered biweekly (Experimental): pTVG-AR (dose: 100 µg) with rhGM-CSF (200 µg). Administered at weeks 0, 2, 12, 14, 24, 26, 36, 38, 48 and 50 (staggered biweekly schedule) for 10 total doses.
  Interventions: Biological: pTVG-AR; Biological: gm-csf

INTERVENTIONS:
Biological: pTVG-AR — Given ID
  Other Names: pTVG-AR vaccine
Biological: gm-csf — Given ID
  Other Names: Recombinant human GM-CSF; rhGM-CSF
  Arms: pTVG-AR with rhGM-CSF biweekly; pTVG-AR with rhGM-CSF staggered biweekly

SUMMARY:
The purpose of this study is to determine if a vaccine called pTVG-AR can enhance the participant's immune response against prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years of age with a histologic diagnosis of adenocarcinoma of the prostate.
* Participant must have metastatic prostate cancer (clinical stage D1 or D2 disease), with previously documented lymph node, soft tissue and/or bone metastases by radiographic imaging (including CT (or MRI) of abdomen and pelvis and bone scintigraphy). Participants in situations in which there is a reasonable clinical suspicion of a second primary tumor (or other non-prostate cancer reason for radiographic abnormalities) are not eligible unless metastatic disease is histologically confirmed to be prostate cancer.
* Participant must have started androgen deprivation therapy (bilateral orchiectomy versus LHRH agonist, and with or without androgen antagonist) at least one month (4 weeks) prior to enrollment and no more than six months (24 weeks) prior to enrollment. Participant must continue the androgen deprivation therapy throughout the study period, and patients are not permitted to change the type of androgen deprivation therapy (e.g. by adding an androgen antagonist) during the course of investigational therapy.
* Participant must have a serum testosterone < 50 ng/dL demonstrated within 1 month of study entry.
* Participant must either not be a candidate for docetaxel chemotherapy for newly diagnosed metastatic prostate cancer, as determined by their treating oncologist, or have declined this therapy
* Participant must have evidence of response to androgen deprivation as defined by a documented decline in serum PSA values from pre-androgen deprivation treatment baseline and without evidence of PSA progression while on androgen deprivation (defined by PCWG2 criteria as a 25% increase in serum PSA and an absolute increase of 2 ng/mL over nadir).
* Participant with a prior history of a second malignancy are eligible provided they have been treated with curative intent and have been free of disease greater than three years. There will be no exclusion for patients with a history of basal cell carcinoma, squamous cell skin cancer, or other in situ carcinoma that has been adequately treated.
* Participant who are sexually active must use a reliable form of contraception while on study and for 4 weeks after the last immunization.
* Eastern Cooperative Oncology Group (ECOG) performance score < 2.
* Participant must have adequate hematologic, renal and liver function as defined by: WBC > 3000/mm3, hematocrit > 30%, platelet count > 100,000/mm3, serum creatinine < 1.6 mg/dl or a calculated creatinine clearance > 60 cc/min, and serum bilirubin < 2.0 mg/dl, within 4 weeks prior to first immunization.
* Participant must be informed of the experimental nature of the study and its potential risks and must sign an IRB-approved written informed consent form indicating such an understanding.

Exclusion Criteria:

* Small cell or other (non-adenocarcinoma) variant prostate cancer histology.
* Participant cannot have evidence of immunosuppression or have been treated with immunosuppressive therapy, such as chemotherapy, chronic treatment dose corticosteroids (greater than the equivalent of 10 mg prednisone per day), or radiation therapy to >30% of the bone marrow, within 6 months of the first vaccination. Treatment or salvage radiation therapy encompassing < 30% of bone marrow must have been completed 4 weeks prior to the first vaccination.
* Seropositive for HIV, hepatitis B (HBV) or hepatitis C (HCV) per participant history.
* Participant previously treated with neoadjuvant and/or adjuvant androgen deprivation (e.g. with radiation therapy) prior to the 6-month eligibility period are allowed, assuming they did not meet criteria for progression (defined by PCWG2 criteria as a 25% increase in serum PSA and an absolute increase of 2 ng/mL over nadir) while on treatment.
* Participant must not be concurrently taking other medications or supplements with known hormonal effects (other than LHRH agonists or non-steroidal anti-androgen), including PC-SPES, megestrol acetate, finasteride, ketoconazole, estradiol, or Saw Palmetto. All other medications with possible anti-cancer effects must be discussed with the Protocol Principal Investigator prior to study entry.
* Participant previously treated with herbal supplements as described in 6.B.5, or other potential or experimental therapies for prostate cancer (apart from LHRH agonists and antiandrogens as described in 6.A.3 above), must have been discontinued these treatments and completed at least a one-month washout prior to first vaccination.
* Participant must not have plans to receive concomitant chemotherapy, other biological or immune therapies, or radiation therapy for the treatment of prostate cancer during the period of study treatment.
* Participant must not have known psychological or sociological conditions, addictive disorders or family problems, which would preclude compliance with the protocol.
* Participant must not have known allergic reactions to GM-CSF or the tetanus vaccine.
* Prior treatment with another experimental anti-tumor vaccine is permissible.
* Participant with unstable or severe intercurrent medical conditions or laboratory abnormalities that would impart, in the judgment of the Protocol Principal Investigator, excess risk associated with study participation or study agent administration.
* Unable or unwilling to undergo two leukapheresis procedures.
* Participant with medical conditions precluding leukapheresis.
* Participant cannot have concurrent enrollment on other phase I, II, or III investigational treatment studies for the treatment of prostate cancer.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-08-24 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2020-11-28 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events following serial intradermal vaccinations of a DNA vaccine encoding AR LBD, with or without GM-CSF as an adjuvant, in patients with metastatic prostate cancer | From first immunization to Week 72
Immune Response Rate | From first immunization to Week 72

SECONDARY OUTCOMES:
Median Progression-Free Survival | From first immunization to Week 72
  Median time to PSA progression will be determined as a function of the date the participant started on androgen deprivation and as a function of treatment start date (week 0). Development of new metastases or discontinuation of study to begin other therapy, while not expected to precede a PSA progression endpoint, would also constitute a progression endpoint.
18-Month Progression-Free Survival | 18 months
The proportion of patients with a T-cell immune response. | From first immunization to Week 72
  Generation of AR LBD-specific peptide-specific CD8+ T cells as defined by ELISPOT and tetramer staining
The number of patients that generate antigen specific tolerance | From first immunization to Week 72
  Antigen-specific tolerance generation following multiple immunizations
Association between pre-existing immune responses to the AR LBD and development of subsequent effector and memory T-cell immune response | From first immunization to Week 72
Association between development of antigen-specific T cells and 18-month progression-free survival | From first immunization to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G. McNeel, M.D., Ph.D., Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (3):
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Washington Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Kyriakopoulos CE, Eickhoff JC, Ferrari AC, Schweizer MT, Wargowski E, Olson BM, McNeel DG. Multicenter Phase I Trial of a DNA Vaccine Encoding the Androgen Receptor Ligand-binding Domain (pTVG-AR, MVI-118) in Patients with Metastatic Prostate Cancer. Clin Cancer Res. 2020 Oct 1;26(19):5162-5171. doi: 10.1158/1078-0432.CCR-20-0945. Epub 2020 Jun 8. PMID 32513836
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/